CLINICAL TRIAL: NCT01616810
Title: Lower Urinary Tract Symptoms Screening Questionnaire Validation STudy
Brief Title: Lower Urinary Tract Symptoms Screening Questionnaire
Acronym: LUTS-2
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 04-227
Record Dates: First submitted 2011-08-26; First posted 2012-06-12 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Cystocele
Keywords: urinary tract
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation: Healthy participants

SUMMARY:
The purpose of this study is to determine the validity of a screening tool which has been designed to detect the presence or absence of lower urinary tract symptoms in the general female population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, 18 years of age and older with any gynecological symptoms

Exclusion Criteria:

* Patients with lower urinary tract symptoms and pelvic floor dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants, 18 years of age and older with any gynecological symptoms other than lower urinary tract symptoms or pelvic floor dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Presence or absence of lower urinary tract symptoms in the general female population | Five years
  To validate the effectiveness of a screening tool in detecting the presence or absence of lower urinary tract symptoms in the general female population.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Soroka, MD, FRCS(C), Principal Investigator — Unity Health Toronto